CLINICAL TRIAL: NCT03607448
Title: Freestyle Libre Flash Glucose Monitoring System Accuracy Study
Brief Title: Freestyle Libre Flash Glucose Monitoring System
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-VAL-18174
Record Dates: First submitted 2018-07-27; First posted 2018-07-31 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Diabetes Mellitus Type 1 and Type 2: Subjects will wear the Abbott Sensor Based Glucose Monitoring Systems and expected to perform at least 8 capillary BG test per day. Site Staff will determine when subject will undergo either a hypoglycemia induction or a hyperglycemia induction. Study staff will perform IV blood draw to obtain blood plasma for YSI sampling every 15 min when glucose as measured by YSI is above 70mg/dL and below 240 mg/dL.
  Interventions: Device: Freestyle Libre Flash Glucose Monitoring System

INTERVENTIONS:
Device: Freestyle Libre Flash Glucose Monitoring System — Subjects will wear the Abbott Sensor based FreeStyle Libre Flash Glucose Monitoring System and will receive no treatment except for safety purposes

SUMMARY:
The purpose of this study is to characterize the Freestyle Libre Flash Glucose Monitoring System performance with respect to YSI reference venous plasma sample measurements.

DETAILED DESCRIPTION:
Up to 200 subjects will be enrolled in this study at a total of 6 clinical research sites in the United States. Subjects will wear a total of two (2) sensors, one on the back of each upper arm. Each Sensor will have a paired Reader that will be given to the subject. All Readers will be masked during the study (i.e. subjects will not be able to view glucose results obtained from the Sensor on the Reader screen). Subjects will be asked to perform at least 8 capillary Blood Glucose (BG) tests per day using the primary Reader. Interstitial glucose readings from each Sensor will be obtained with the corresponding Readers immediately following each BG test. Subjects will be instructed to report any problems with the device. Subjects will make six (6) scheduled visits to the clinical study site, including the Enrollment/Screening Visit (Visit 1). Subjects will have three (3) in-clinic visits during which intravenous blood draws and YSI reference testing will occur.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject must have type 1 or type 2 diabetes.
* Subject must require insulin therapy through an insulin pump and/or multiple daily insulin injections (at least 3 injections daily).
* Willing to perform a minimum of 8 finger sticks per day while wearing the sensor in the study.
* Subject must be able to read and understand English.
* Willing to have their blood sugar manipulated during in-clinic sessions.
* In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
* At the time of enrollment, subject must be available to participate in all study visits.
* Subject must be willing and able to provide written signed and dated informed consent.
* Additional criteria for hypoglycemia induction.
* Known insulin sensitivity factor.

Exclusion Criteria:

* Subject has a history of hypoglycemia unawareness.
* Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
* Subject is pregnant, attempting to conceive or not willing and able to practice birth control during the study duration (applicable to female subjects only).
* Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
* Subject has had an episode of severe hypoglycemia requiring intervention from a health care professional (i.e. EMT assistance, emergency room visit, or hospital admission) within the last three (3) months.
* Subject is currently participating in another clinical trial.
* Subject has donated blood within 112 days (3.7 months) prior to the beginning of the study activities.
* Subject has both hemoglobin (Hb) and hematocrit levels that are 10% or more below the normal ranges (For reference low end of the normal range for Hb for males is 14 g/dL and for females is 12 g/dL; low end of the normal hematocrit is 40% for men and 36% for women).
* Subject has concomitant medical condition which, in the opinion of the investigator, could present a risk to the safety or welfare of the subject or study staff. Such conditions include but are not limited to:
* History of HIV, Hepatitis B or C
* Subject has X-ray, MRI, CT or diathermy appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
* Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Type 1 or Type 2 diabetes requiring multiple daily insulin injections (MDI) or continuous subcutaneous insulin infusion (CSII).
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
System Performance | approximately 45 days
  System Performance will be characterized with respect to YSI reference venous plasma measurements

SECONDARY OUTCOMES:
System Related Adverse Device Effects | Up to 45 days
  System will be characterized by Adverse Device Effects and Serious Adverse Device Effects experienced by study participants

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara Karinka, PhD, Study Director — Abbott Diabetes Care
Locations (5):
- United States (5):
  - AMCR, Escondido, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Diablo Clinical Research, Walnut Creek, California
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Rainier Clinical Research Center, Renton, Washington

REFERENCES:
- [Derived] Alva S, Bailey T, Brazg R, Budiman ES, Castorino K, Christiansen MP, Forlenza G, Kipnes M, Liljenquist DR, Liu H. Accuracy of a 14-Day Factory-Calibrated Continuous Glucose Monitoring System With Advanced Algorithm in Pediatric and Adult Population With Diabetes. J Diabetes Sci Technol. 2022 Jan;16(1):70-77. doi: 10.1177/1932296820958754. Epub 2020 Sep 19. PMID 32954812